CLINICAL TRIAL: NCT06783335
Title: The Real-World Effectiveness of The Cordella Pulmonary Artery Sensor System in Patients With Chronic Heart Failure: A Comparative Analysis to Standard of Care Pharmacologic Therapy
Brief Title: Real World Effectiveness of the Cordella Pulmonary Artery Sensor System in Patients With Chronic Heart Heart Failure
Acronym: LOWER-PAP
Status: Recruiting | Type: Observational
Sponsor: Endotronix, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: OS-2025-001
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure NYHA Class III; Heart Failure
Keywords: Heart failure; Heart Disease; Pulmonary Artery Pressure Sensor; Cardiovascular Disease; Cordella
MeSH Terms: conditions — Heart Failure; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Cordella PA Sensor System — * Patients who receive the Cordella PA Sensor System for monitoring chronic heart failure
  * These patients will be monitored for 2 years after receiving the device
  * Patients must be on guideline-directed medical therapy appropriate for their ejection fraction status
Drug: Standard of Care Pharmacologic Therapy — * Patients with chronic heart failure who receive standard medical care without PA pressure monitoring
  * These patients will be monitored for 2 years
  * Patients must be on guideline-directed medical therapy appropriate for their ejection fraction status

SUMMARY:
This retrospective, non-randomized cohort study will evaluate how well the Cordella PA Sensor System works compared to standard medication treatment in people with chronic heart failure. The study will track patients for two years to see if those using the Cordella system have fewer deaths and hospitalizations related to heart failure.

DETAILED DESCRIPTION:
The study will compare two groups of patients with chronic heart failure:

* One group will use the Cordella PA Sensor System, which monitors heart pressure from home
* The other group will receive standard heart failure medications without a pressure monitoring system

The main goal is to see if patients using the Cordella system have fewer heart failure-related hospital stays and a lower death rate over a two-year period. The study will look especially closely at results for:

* Men and women separately
* Patients with different types of heart failure (preserved or reduced heart function)
* Patients aged 75 and older
* Different racial and ethnic groups
* Patients with kidney disease
* Patients with existing heart devices

The study will use real-world data from:

* Patients using the Cordella system in routine medical care
* Similar patients receiving standard care, identified through medical records and insurance claims Both groups of patients will be carefully matched to ensure they are similar in age, gender, and other important factors that could affect the results.

ELIGIBILITY:
Inclusion Criteria for Cordella PA Sensor System Cohort:

* Received Cordella PA Sensor System implant between 10/1/2024-12/31/2029
* Documented chronic heart failure with NYHA Class III symptoms
* On guideline-directed medical therapy based on ejection fraction status:

  * For reduced EF (≤40%): At least one fill of ACE/ARB/ARNI, MRA, BB, or SGLT2i, and one fill of a loop diuretic
  * For preserved EF (>40%): At least one fill of a loop diuretic
* Has continuous health insurance enrollment for 12 months prior to implant

Inclusion Criteria for Standard of Care Control Cohort:

* Two or more encounters with diagnosis codes for chronic systolic and/or diastolic heart failure
* Documented ejection fraction reading within 6 months (+ or -) of second heart failure encounter
* On guideline-directed medical therapy based on ejection fraction status:

  * For reduced EF (≤40%): At least one fill of ACE/ARB/ARNI, MRA, BB, or SGLT2i, and one fill of a loop diuretic
  * For preserved EF (>40%): At least one fill of a loop diuretic
* Has continuous health insurance enrollment for 12 months prior to study entry

Exclusion Criteria:

* No implanted pulmonary artery sensor or monitoring at any time (Standard of Care Control Cohort only)
* Record of temporary mechanical circulatory support during baseline period
* Diagnosis of cardiogenic shock during baseline period
* Receiving palliative care/hospice during baseline period
* Record of end-stage renal disease during baseline period
* Unable to take dual antiplatelet therapy or anticoagulants for one month post implant (Cordella Cohort only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NYHA III chronic HF
Sampling Method: Non-Probability Sample
Enrollment: 2150 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite of All-cause Mortality and Heart Failure Hospitalizations | up to 24 months
  * Description: The cumulative number of all-cause deaths and heart failure hospitalizations
  * Time Frame: 2 years after study entry (time zero)
  * Statistical Analysis Plan: The primary analysis will use an Andersen-Gill recurrent event model to account for multiple hospitalizations within individuals
  * Primary outcome will be assessed in the overall population

SECONDARY OUTCOMES:
Composite Outcome in Racial and Ethnic Subgroups | up to 24 months
  The cumulative number of all-cause deaths and heart failure hospitalizations in:
  * Black/African American patients
  * Asian patients
  * Hispanic patients
Composite Outcome in Patients with Chronic Kidney Disease | up to 24 months
  The cumulative number of all-cause deaths and heart failure hospitalizations in patients with documented chronic kidney disease
Composite Outcome in Patients with Cardiac Devices | up to 24 months
  The cumulative number of all-cause deaths and heart failure hospitalizations in patients with indwelling cardiac implantable electronic devices
Composite Outcome in Patients by Ejection Fraction | up to 24 months
  The cumulative number of all-cause deaths and heart failure hospitalizations in patients with HF with reduced ejection fraction and patients with HF with preserved ejection fraction
Composite Outcome in Patients Age 75+ | up to 24 months
  The cumulative number of all-cause deaths and heart failure hospitalizations in patients age 75+

CONTACTS AND LOCATIONS:
Overall Officials: Joanna VanHouten, PhD, Principal Investigator — Endotronix, Inc.
Locations (1):
- Endotronix, Naperville, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
This study will leverage de-identified data sourced from Optum which has limits on sharing its proprietary data.